CLINICAL TRIAL: NCT03125005
Title: Accuracy of Methemoglobin Measurement for Rainbow Universal Pulse Oximeter Sensor
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Masimo Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: TR22640-BICK0001
Record Dates: First submitted 2017-04-14; First posted 2017-04-24 (Actual); Results first posted 2017-06-06 (Actual); Last update posted 2017-07-27 (Actual); Status verified 2017-06

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Rainbow Universal Pulse Oximeter Sensor (Experimental): All subjects will be enrolled in the test group and will receive Rainbow Universal Pulse Oximeter Sensor.
  Interventions: Device: Rainbow Universal Pulse Oximeter Sensor

INTERVENTIONS:
Device: Rainbow Universal Pulse Oximeter Sensor

SUMMARY:
In this study, the level of methemoglobin (HbMet) will be increased in a controlled manner by administering sodium nitrite intravenously in healthy volunteers. The accuracy of a noninvasive HbMet sensor will be assessed by comparison to blood measurements from a laboratory analyzer.

ELIGIBILITY:
Inclusion Criteria

* The subject is male or female, aged ≥18 and <50.
* The subject is in good general health with no evidence of any medical problems.
* The subject is fluent in both written and spoken English.
* The subject has provided informed consent and is willing to comply with the study procedures.

Exclusion Criteria:

* The subject is obese (BMI>30).
* The subject has a known history of heart disease, lung disease, kidney or liver disease.
* Diagnosis of asthma, sleep apnea, or use of CPAP.
* Subject has diabetes.
* Subject has a clotting disorder.
* The subject has a hemoglobinopathy or history of anemia, per subject report or the first blood sample, that in the opinion of the investigator, would make them unsuitable for study participation.
* The subject has any other serious systemic illness.
* The subject is a current smoker.
* Any injury, deformity, or abnormality at the sensor sites that in the opinion of the investigators' would interfere with the sensors working correctly.
* The subject has a history of fainting or vasovagal response.
* The subject has a history of sensitivity to local anesthesia or allergy to the study drugs.
* The subject has a diagnosis of Raynaud's disease.
* The subject has unacceptable collateral circulation based on exam by the investigator (Allen's test).
* The subject is pregnant, lactating or trying to get pregnant.
* The subject has a history of migraine headaches.
* The subject is currently taking antidepressants.
* The subject is unable or unwilling to provide informed consent, or is unable or unwilling to comply with study procedures.
* The subject has any other condition, which in the opinion of the investigators' would make them unsuitable for the study.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 51 (Actual)
Dates: Start 2012-04-12 (Actual); Primary Completion 2012-06-21 (Actual); Study Completion 2012-06-21 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Masimo Clinical Lab, Irvine, California
  - University of San Francisco, San Francisco, California

RESULTS

PARTICIPANT FLOW:
Groups:
- Rainbow Universal Pulse Oximeter Sensor: All subjects will be enrolled in the test group and will receive Rainbow Universal Pulse Oximeter Sensor.
  Rainbow Universal Pulse Oximeter Sensor
Period: Overall Study
Arm/Group | Rainbow Universal Pulse Oximeter Sensor
Started | 51
Completed | 51
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Rainbow Universal Pulse Oximeter Sensor
Number analyzed (Participants) | 51
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 51
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29
  Male | 22
Region of Enrollment [Number; unit: participants]
  United States | 51

OUTCOME MEASURES:

1. Primary Outcome: Accuracy of Sensor by Arms Calculation
Description: Accuracy willl be determined by comparing the noninvasive blood methemoglobin measurement (expressed as a percentage of total hemoglobin) of the pulse oximeter to that obtained from a blood sample and calculating the arithmetic root mean square(Arms) error value.
Time Frame: 5 hours
Measure: Number; unit: Percentage of total hemoglobin
Arm/Group | Rainbow Universal Pulse Oximeter Sensor
Number analyzed (Participants) | 51
Percentage of total hemoglobin | 0.63

ADVERSE EVENTS:
Arm/Group | Rainbow Universal Pulse Oximeter Sensor
All-Cause Mortality (participants affected / at risk) | 0/51
Serious Adverse Events (participants affected / at risk) | 0/51
Other Adverse Events (participants affected / at risk) | 0/51

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less